CLINICAL TRIAL: NCT06498063
Title: Renal Extraction of Glucagon and Renal Effects of Glucagon
Brief Title: The Underlying Mechanisms Regarding the Effect of Glucagon on the Kidneys Will be Investigated in Healthy Males.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ali Asmar (Other)
Collaborators: University of Copenhagen (Other); The Augustinus Foundation, Denmark. (Other); The Novo Nordic Foundation (Other)
Responsible Party: Sponsor-Investigator, Ali Asmar, Chief Physician, Associate Professor, PhD, MD, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-22019483; 20-1914; 21-1518 (Other Grant/Funding Number: Augustinus Fonden); NNF21OC0070308 (Other Grant/Funding Number: Novo Nordisk Fonden)
Record Dates: First submitted 2024-02-22; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — Glucagon; exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Glucagon (Experimental): Glucagon infusion of 5 ng·kg-1·min-1 from 0-60 minutes and 10 ng·kg-1 ·min-1 from 60-120 minutes.
  Interventions: Other: Glucagon; Other: Placebo; Other: Glucagon and exendin 9-39
- Glucagon+Exendin9-39 (Experimental): Glucagon (infusion of 5 ng·kg-1·min-1 from 0-60 minutes) and glucagon (infusion of 10 ng·kg-1 ·min-1 from 60-120 minutes) + a GLP-1R antagonist, exendin 9-39 (900 pmol·kg-1·min-1 from -30-120 minutes).
  Interventions: Other: Glucagon; Other: Placebo; Other: Glucagon and exendin 9-39
- Sodium chloride (Placebo comparator) (Placebo Comparator): NaCl (0.9%)
  Interventions: Other: Glucagon; Other: Placebo; Other: Glucagon and exendin 9-39

INTERVENTIONS:
Other: Glucagon — Glucagon infusion of 5 ng·kg-1·min-1 from 0-60 minutes and 10 ng·kg-1 ·min-1 from 60-120 minutes.
Other: Placebo — Placebo (0.9% NaCl).
Other: Glucagon and exendin 9-39 — Glucagon (infusion of 5 ng·kg-1·min-1 from 0-60 minutes) and glucagon (infusion of 10 ng·kg-1 ·min-1 from 60-120 minutes) + a GLP-1R antagonist, exendin 9-39 (900 pmol·kg-1·min-1 from -30-120 minutes).

SUMMARY:
The goal of this crossover study is to investigate to what extend glucagon affects the kidneys. The main questions it aims to answer are:

Does glucagon regulate kidney function through extraction in the kidney in addition to glomerular filtration? Does glucagon regulate kidney function by increasing renal plasma flow and glomerular filtration rate? Does glucagon regulate kidney function by increasing renal salt excretion?

DETAILED DESCRIPTION:
In patients with type 2 diabetes mellitus, plasma concentrations of glucagon are inappropriately high (hyperglucagonemia). Hyperglucagonemia has been speculated to contribute to the pathophysiology of diabetic kidney disease. Previously, glucagon has been assumed to cause glomerular hyperfiltration associated with urinary excretion of small proteins, a characteristic of early type 2 diabetic kidney injury. Further, glucagon has been shown to acutely increase urinary excretion of urea, sodium, and potassium, and patients with end-stage renal disease have elevated plasma levels of glucagon.

The purpose of this study is to clarify the underlying mechanisms behind the physiological effects of glucagon on kidney function and the kidney's ability to clear glucagon from the blood in healthy males. Specifically, the investigators aim to answer the following questions:

Does glucagon regulate kidney function through extraction in the kidney in addition to glomerular filtration? Does glucagon regulate kidney function by increasing renal plasma flow and glomerular filtration rate? Does glucagon regulate kidney function by increasing renal salt excretion?

The renal extraction of glucagon and the renal effects of glucagon will be investigated during a constant glucagon infusion in 10 healthy men aged 20-60 years. The study will be placebo-controlled. Each subject will participate in three independent and randomized trial days with a washout period of at least four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-60 years
* Normal health ascertained through questioning and medical examination
* Normal values for blood concentrations of fasting plasma glucose, fasting plasma total cholesterol, fasting triglycerides, HDL, LDL, creatinine, liver function, and electrolytes
* Informed consent

Exclusion Criteria:

* Immunosuppressive treatment in the preceding 12 months
* Alcohol abuse
* Medical treatment with oral glucocorticoids, dipeptidyl peptidase-4 (DPP-4) inhibitors, or GLP-1 receptor agonists, which, in the opinion of the investigator, may interfere with glucose metabolism
* Use of lithium
* Medical treatment that affects insulin secretion or cardiovascular performance measures
* Liver disease (ALT > 2x normal value)
* Renal impairment (se-creatinine > 130 μM and/or albuminuria)

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-03-28 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Natriuresis | Analyzed from urine samples at -60, 0, 60 and 120 minutes
  From urine samples, unit mmol/L
Glucagon extraction | Analyzed from blood samples drawn at -30, 0, 20, 40, 60, 80, 100, 120, 140, 160 and 180 minutes
  From blood samples, unit pmol/L

SECONDARY OUTCOMES:
Glomerular filtration rate | Measured via Fick's principle during steady state using [99mTc]Tc-DTPA (diethylene-triamine-pentaacetate) as a tracer given as a constant infusion from -210 to 180 min.
  Unit mL/min
Diuresis | Analyzed from urine samples at -60, 0, 60 and 120 minutes
  from urine samples, unit mL/min
Renal Blood Flow | Measured via Fick's principle during steady state using [99mTc]Tc-DTPA (diethylene-triamine-pentaacetate) as a tracer given as a constant infusion from -210 to 180 min.
  Unit mL/min
Urea | Analyzed from blood samples drawn at -30, 0, 20, 40, 60, 80, 100, 120, 140, 160 and 180 minutes
  Unit mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Ali Asmar, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Physiological laboratory, Bispebjerg Hospital, Research Unit, Clinical Physiology / Nuclear Medicine Department, Copenhagen, Denmark